CLINICAL TRIAL: NCT03895034
Title: A Single Center Exploratory Study to Evaluate the Use of the RxSight Light Adjustable Lens (LAL) and the Light Delivery Device (LDD) to Improve Visual Outcomes
Brief Title: Exploratory Study to Evaluate the Use of the RxSight Light Adjustable Lens (LAL) and the Light Delivery Device (LDD) to Improve Visual Outcomes
Status: Completed | Type: Interventional
Sponsor: RxSight, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-032
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Results first posted 2021-09-22 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-04

CONDITIONS: Aphakia; Cataract
Keywords: Light Adjustable Lens; Intraocular lens; LAL
MeSH Terms: conditions — Aphakia; Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- Light adjustable lens (LAL) and Light Delivery Device (LDD) (Experimental)
  Interventions: Device: Light Adjustable lens (LAL) and Light Delivery Device (LDD)

INTERVENTIONS:
Device: Light Adjustable lens (LAL) and Light Delivery Device (LDD) — Eligible eyes will receive Light adjustable lens with Light delivery Device treatments

SUMMARY:
The objective of this study is to evaluate, for the visual correction of aphakia, whether the RxSight Light Adjustable Lens (LAL) and Light Delivery Device (LDD) can be used to improve visual outcomes after performing adjustments of the LAL with the LDD. This is an exploratory study. No primary effectiveness endpoints will be identified.

ELIGIBILITY:
Inclusion Criteria:

* Must sign a written Informed Consent form and be willing to undergo cataract surgery for unilateral or bilateral implantation of the RxLAL.
* Between the ages of 40 and 80 inclusive on the day the cataract surgery is performed.
* Study eye must have cataract causing reduction in best corrected distance visual acuity (BCDVA) to a level of 20/32 or worse with or without a glare source.
* Willing and able to comply with the requirements for study specific procedures and visits.

Exclusion Criteria:

* Study eye with pseudoexfoliation.
* Study eye with diabetes with any evidence of retinopathy.
* Study eye with evidence of glaucomatous optic neuropathy.
* Study eye with history of uveitis.
* Study eye with prior history of Intacs, Radial keratotomy (RK), Conductive keratoplasty (CK), Astigmatic keratotomy (AK), Phakic Implantable Collamer Lens (ICL), Corneal Inlay, or with previous pterygium excision unless the pterygium did not extend more than 2mm onto the cornea from the limbus.
* Subjects taking systemic medication that may increase sensitivity to UV light.
* Subjects taking a systemic medication that is considered toxic to the retina such as tamoxifen.
* Study eye with history of ocular herpes simplex virus.
* Study eye with history of a congenital color vision defect

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CODET Vision Institute, Tijuana, Mexico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD)
Started | 66; 111 Eyes
Completed | 64; 109 Eyes
Not Completed | 2; 2 Eyes
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD)
Number analyzed (Participants) | 66
Number analyzed (Eyes) | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 66
  White | 0
  Black | 0
  Other | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 66
Eyes [Count of Units; unit: Eyes]
  OD | 56
  OS | 55

OUTCOME MEASURES:

1. Primary Outcome: Percent of Eyes With Uncorrected Distance Visual Acuity (UCDVA) of 20/20 or Better
Time Frame: 3 months post op
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD)
Number analyzed (Participants) | 66
Number analyzed (Eyes) | 109
Eyes | 101

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 3 months
Description: The at Risk number in All-Cause Mortality represent whole participants while the at Risk number in the Serious and Other (Not Including Serious) Adverse Events tables represent the number of eyes. Non-ocular adverse events were not collected.
Arm/Group | Light Adjustable Lens (LAL) and Light Delivery Device (LDD)
All-Cause Mortality (participants affected / at risk) | 0/66
Serious Adverse Events (participants affected / at risk) | 0/111
Other Adverse Events (participants affected / at risk) | 25/111
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Light Adjustable Lens (LAL) and Light Delivery Device (LDD) (N=111)
Anterior Capsule Rupture (Eye disorders) | 1 (1)
BCDVA Drop of 10 letters of more (Eye disorders) | 1 (2)
Corneal Erosion (Eye disorders) | 1 (1)
Corneal Guttata (Eye disorders) | 2 (2)
Cystoid Macular Edema (Eye disorders) | 1 (1)
Iris Atrophy (Eye disorders) | 1 (1)
Iritis (Eye disorders) | 3 (4)
Posterior Capsular Opacity (Eye disorders) | 2 (2)
Superficial Punctate Keratitis (Eye disorders) | 11 (11)
Vision changes including night vision changes (Eye disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT03895034/Prot_SAP_000.pdf